CLINICAL TRIAL: NCT03172390
Title: In Vivo Evaluation of Growth and Risk of Rupture of Dilated Ascending Aorta Using 4D Cardiac Magnetic Resonance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1708028; 2017-A00871-52 (Other: ANSM)
Record Dates: First submitted 2017-05-23; First posted 2017-06-01 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Aortic Rupture
Keywords: Ascending aorta aneurysm; Aortic wall shear stress; 4D phase contrast Cardiovascular Magnetic Resonance; Aortic dissection
MeSH Terms: conditions — Aortic Rupture; Aneurysm, Ascending Aorta; Aortic Dissection

STUDY DESIGN:
Intervention Model Description: Prospective cohort
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort of patients : ascending aorta dilatation (Experimental): measure of ascending aorta quality and quantity parameters by 4D Cardiac magnetic resonance
  Interventions: Device: 4D Cardiac Magnetic Resonance

INTERVENTIONS:
Device: 4D Cardiac Magnetic Resonance — 4D Cardiac Magnetic Resonance for patients with a ascending aorta dilatation without current indication for surgery for measured parameters of ascending aorta

SUMMARY:
Ascending aorta aneurysmal disease is common and can be complicated by dissection or rupture. There is substantial variation in individual aneurysm progression: established risk factors for an accelerated aneurysm growth rate include initial size or localization, the presence of aortic valve disease, congenital bicuspid aortic valve or connective tissue disorders.

DETAILED DESCRIPTION:
Although there is an increased lifetime risk when the aortic diameter exceeds 6 cm, predicting aneurysm progression is nearly impossible and dissection and rupture also occur at diameters under 6 cm. The assessment of aortic hemodynamics and the presence of altered flow patterns, as well as distribution and changes in wall shear stress (WSS) and the oscillatory shear index (OSI), using 4D phase contrast cardiovascular magnetic resonance (CMR) may provide further insights in how aneurysms develop and in assessing the risk of dissection. The purpose of this study was to investigate in patients with dilated ascending aorta the flow patterns and vessel wall parameters in order to correlate these hemodynamics factors with changes in aorta size.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Supra-coronary aortic diameter measured by CT-scan or transthoracic/trans-esophageal echocardiography between 40 and 45 mm in case of presence of aortic valve disease, bicuspid aortic valve or connective tissue disease and between 40 and 50 mm in case of absence of aortic valve disease, bicuspid aortic valve disease or connective tissue.
* Informed consent for participation in the study

Exclusion Criteria:

* Contraindication to MRI
* Patient's refusal to participate in the study and / or inability to express agreement or signing the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
Correlation between wall shear stress (WSS) and aorta diameter in patient with dilated ascending aorta | From baseline to 1 year
  Aorta diameter [mm] is assessed by 4D phase contrast cardiovascular magnetic resonance (CMR) Wall shear stress (WSS) in aorta [Pa] is assessed by 4D phase contrast cardiovascular magnetic resonance (CMR).

SECONDARY OUTCOMES:
Aorta parameters associated with change in aorta diameter | From baseline to 1 year
  Aorta parameters are a composite outcome :
  * the oscillatory shear index (OSI)
  * pulse wave velocity=PWV [m/s] assessed by 4D phase contrast cardiovascular magnetic resonance (CMR). Aorta diameter [mm] is assessed by 4D phase contrast cardiovascular magnetic resonance (CMR)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Saint-Etienne, Saint-Étienne-de-Montluc, Pays de la Loire Region, France

IPD SHARING:
Plan to Share IPD: No